CLINICAL TRIAL: NCT01654965
Title: A Phase I Study of ARQ 197 in Combination With IV Topotecan in Advanced Solid Tumors With an Expansion Cohort in Small Cell Lung Cancer
Brief Title: Tivantinib and Topotecan Hydrochloride in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01220; NCI-2012-01220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000738072; PHI-68; PHI-68 (Other: City of Hope Comprehensive Cancer Center); 9152 (Other: CTEP); P30CA033572 (NIH); U01CA062505 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — pegfilgrastim; ARQ 197; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (tivantinib, topotecan hydrochloride, pegfilgrastim) (Experimental): Patients receive tivantinib PO BID on days 1-21, topotecan hydrochloride IV over 30 minutes on days 1-5, and pegfilgrastim SC on day 6. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pegfilgrastim; Other: Pharmacological Study; Drug: Tivantinib; Drug: Topotecan Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; HSP-130; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF
Other: Pharmacological Study — Correlative studies
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)

SUMMARY:
This phase I trial studies the side effects and best dose of tivantinib and topotecan hydrochloride in treating patients with advanced or metastatic solid tumors. Tivantinib and topotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended phase 2 dose (RP2D) for the combination of ARQ 197 (tivantinib) and intravenous (IV) topotecan (topotecan hydrochloride).

II. To describe the toxicities of ARQ 197 and IV topotecan at each dose studied.

III. To characterize the pharmacokinetic behavior of ARQ 197 given concurrent use of IV topotecan.

IV. To document all clinical responses to ARQ 197 with IV topotecan.

OUTLINE: This is a dose-escalation study of tivantinib and topotecan hydrochloride.

Patients receive tivantinib orally (PO) twice daily (BID) on days 1-21, topotecan hydrochloride IV over 30 minutes on days 1-5, and pegfilgrastim subcutaneously (SC) on day 6. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; for the expansion group, patients must have histologically or cytologically confirmed small cell lung cancer previously treated with one or more chemotherapy or chemoradiotherapy regimens, at least one of which must have been platinum-based

  * As of amendment dated 01/24/2014 the study will not be pursuing an expansion cohort in small cell lung cancer
* Karnofsky >= 60%
* Life expectancy of greater than 12 weeks
* Hemoglobin >= 9.0 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (=< 5 X institutional upper limit of normal if the rise can be attributed to liver metastases)
* Serum creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ARQ 197 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with untreated brain metastases should be excluded from this clinical trial; however patients with stable brain disease (off corticosteroids) at least 2 weeks after completion of appropriate therapy for their brain metastases are eligible; patients who require enzyme-inducing anti-convulsants (EIAC) should be switched to non-EIAC and be on a stable dose of the new agent for at least 2 weeks prior to treatment on this protocol
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197 or topotecan
* The metabolism and consequently overall pharmacokinetics of ARQ 197 could be altered by inhibitors and/or inducers or other substrates of cytochrome P450 2C19 (CYP2C19) and cytochrome P450 3A4 (CYP3A4); while inhibitors/inducers of these cytochrome P450 isoenzymes are not specifically excluded, investigators should be aware that ARQ 197 exposure may be altered by the concomitant administration of these drugs; caution should be applied when CYP2C19 inhibitors such as omeprazole, fluvoxamine, fluconazole, ticlopidine, rabeprazole, fluoxetine, and moclobemide, or strong CYP3A4 inhibitors such as atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, ciprofloxacin, telithromycin, troleandomycin (TAO), or voriconazole, are used as concomitant therapy; because the lists of these agents are changing, it is important to consult an updated list; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* History of congestive heart failure defined as class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as >= grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ARQ 197
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients previously treated with topotecan are ineligible
* Patients previously treated with ARQ 197 are ineligible
* Patients unable to swallow ARQ 197 pills are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events graded according to the NCI CTCAE version 4.0 | Up to 4 weeks
  The toxicities observed at each dose level will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by CTCAE), attribution, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.

SECONDARY OUTCOMES:
Tumor response as evaluated by Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 4 weeks
  All responses will be reported; because of the potential heterogeneity of the patients, no attempt will be made to summarize these for the patients included in the dose escalation phase.
Progression-free survival (PFS) | The time from start of treatment until first evidence of disease progression or death due to any cause, assessed up to 4 weeks
  PFS will be reported; because of the potential heterogeneity of the patients, no attempt will be made to summarize these for the patients included in the dose escalation phase.
Overall survival (OS) | The time from start of treatment until death due to any cause, assessed up to 4 weeks
  OS will be reported; because of the potential heterogeneity of the patients, no attempt will be made to summarize these for the patients included in the dose escalation phase.

OTHER OUTCOMES:
Pharmacokinetics behavior of tivantinib given concurrently with topotecan hydrochloride | At baseline, at 2, 3, 4, and 8 hours of day 1 and at 12 hours after evening dose of day 4 (on day 5)
  Summarized by dose level with simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations (if numbers and distribution permit). Scatterplots will be used to explore possible associations between the dose and day 1 AUC, dose and levels on day 1 and day 5, and between these pharmacokinetic determinations and toxicity experienced (as reflected in the maximum grade of toxicity experienced). All data summaries based on pharmacokinetic studies will be descriptive and exploratory.
CYP2C19 genotype | Baseline
  The association between CYP2C19 genotype and ARQ 197 levels, and toxicity will also be displayed and summarized. All data summaries based on pharmacodynamic studies will be descriptive and exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania